CLINICAL TRIAL: NCT02112695
Title: Opioid System Cerebral Activity in Endurance Sportswomen - Addiction or Denutrition ? [11C]Diprenorphine PET Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Saint Etienne (Other)
Collaborators: Ministry of Health, France (Other Government)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 1208051; 2013-004733-32 (EudraCT Number)
Record Dates: First submitted 2014-04-10; First posted 2014-04-14 (Estimated); Last update posted 2018-10-29 (Actual); Status verified 2017-10

CONDITIONS: Sports Nutritional Sciences
Keywords: endurance sportswomen; addiction; undernutrition; [11C]diprenorphine Pet; pituitary region
MeSH Terms: conditions — Behavior, Addictive; Malnutrition

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- sportswomen (Experimental): 3 micrograms [11C]diprenorphine
  Interventions: Other: [11C]diprenorphine
- control subjects (Experimental): 3 micrgrams [11C]diprenorphine
  Interventions: Other: [11C]diprenorphine

INTERVENTIONS:
Other: [11C]diprenorphine — 3 micrograms [11C]diprenorphine - intravenous use - 1 time
  Other Names: radiopharmacentical precursor solution

SUMMARY:
Abnormal opioid system have been identified in addictive behavior and activity of the opioid system has also shown a strong link with the nutritional balance. A significant increase in endorphin levels was noticed after exercise, proportional to the duration and intensity of this activity. One brain imaging study showed an increase in opioid activity in athletes after endurance training. However , a decrease in opioid tone related to receptor desensitization in the brain has been raised in the sport and it is possible to feel like , the subject must perform physical exercise more frequently . Consequently, in order to deepen the hypothesis of addiction in high-level sport , the brain opioid activity should be assessed pre- training compared to a group of sedentary control subjects .

Preliminary results of a previous study the investigators are conducting on anorexia nervosa (AN ) show abnormalities that appear to be involved in self addiction anorexia nervosa and the regulation of gonadal function. However, the relation of cause and effect between these anomalies and undernutrition remains to be determined . Given the addictive component in the endurance sport and the variability of the nutritional status of its practitioners , evaluation of brain activity in these subjects could provide additional answers.

ELIGIBILITY:
Inclusion Criteria:

For High-level sportswomen :

* 18-35-year-old
* High-level sportswomen
* BMI>19kg/m2
* Absence of eating disorders
* In pre-competition period
* Signature of written consent

For controls :

* 18-35-year-old
* Sedentary normal weight women
* BMI>19kg/m2
* Normal nutritional markers
* Absence of eating disorders or other psychiatric or organic diseases

Exclusion Criteria:

* Oral contraception
* Heart failure
* Neuroleptics, antiparkinson drugs, alpha-methyl-dopa, beta blockers, inhibitors of monoamine oxidase-A or MOA-B, tricyclic antidepressants, selective serotonin reuptake inhibitor, thyme-regulators (lithium), anticonvulsant drugs, codeine, morphine, drugs containing tramadol, dopaminergic drugs

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 35 (Actual)
Dates: Start 2014-09-15 (Actual); Primary Completion 2017-07-06 (Actual); Study Completion 2017-07-07 (Actual)

PRIMARY OUTCOMES:
[11C]diprenorphine binding potential | 2 weeks
  Value of [11C]diprenorphin binding potential in predifined brains regions. [11C]diprenorphin BP will be evaluated by brain positron emission tomography and MRI exam

SECONDARY OUTCOMES:
correlation [11C]diprenorphine BP | 2 weeks
  Correlation between [11C]Diprenorphine binding potential and plasma endogenous opioid levels
correlation [11C]diprenorphine BP | 2 weeks
  Correlation between [11C]Diprenorphine binding potential and psychometric score evaluating addictive behavior, reward and positive reinforcement
correlation [11C]diprenorphine BP | 2 weeks
  Correlation between [11C]Diprenorphine binding potential and appetite regulating hormones
correlation [11C]diprenorphine BP | 2 weeks
  Correlation between [11C]Diprenorphine binding potential and LH response during GnRH test

CONTACTS AND LOCATIONS:
Overall Officials: Bruno Estour, PU-PH, Principal Investigator — CHU SAINT-ETIENNE
Locations (1):
- Service d'Endocrinologie - CHU Saint-Etienne, Saint-Etienne, France

IPD SHARING:
Plan to Share IPD: No